CLINICAL TRIAL: NCT06925256
Title: Considerin Peripheral Nerve Injury, Is It Safe to Perform Transradial Angiography?
Brief Title: Considering Peripheral Nerve Injury, Is It Safe to Perform Transradial Angiography?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Taner Dandinoğlu, PM&R physician, Bursa City Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2025-PMR-1
Record Dates: First submitted 2025-03-25; First posted 2025-04-13 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Neuropathic Peripheral Pain
Keywords: Nerve Conduction Studies; Nerve damage; Transradial angiography
MeSH Terms: interventions — Nerve Conduction Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with transradial angiography (Experimental): all patients involved evaluated with NCS
  Interventions: Diagnostic Test: nerve conduction study

INTERVENTIONS:
Diagnostic Test: nerve conduction study — median ulnar and radial motor- sensory nerve conduction studies will be performed.

SUMMARY:
So far, apart from a limited number of case reports and small-scale studies, the frequency and severity of this complication have not been objectively evaluated using electromyography (EMG). In this study, presence, severity, and extent of nerve injury (one of the potential complications following the transradial approach (TRA)) were evaluated by EMG studies in patients managed at Bursa City Hospital.

DETAILED DESCRIPTION:
Evaluation of peripheral nerve injury after transradial angiography with nerve conduction studies.

ELIGIBILITY:
Inclusion Criteria:

20-60 years old patiens who applied trans angiograhy were included to study

Exclusion Criteria:

* Having cognitive disorders
* Patients who have story of cardiac pace / ICD,
* History of polyneuropathy,
* Previous nerve damages,
* Deformities on arm,
* Plexopathy,
* Radiculopathy,
* Spinal surgery.
* Having medical treatment for any kind of neuropathy
* Having Cognitive disorders

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Nerve conduction studies (NCS) | 1 day
  NCS (Nerve conduction study) findings obtained after radial intervention A NCS test measures how fast an electrical impulse moves through your nerve. NCS can identify nerve damage. During the test, your nerve is stimulated, often with electrode patches put on your skin. Two electrodes are placed on the skin over your nerve or over a muscle. One electrode stimulates your nerve with a very mild electrical impulse. The other electrode records it. The resulting electrical activity is recorded by another electrode. This is repeated for each nerve being tested. After test below values are obtained;
  * Velocity (meter/second),
  * Action potential amplitude (miliVolt)
  * Onset latans (milisecond)

IPD SHARING:
Plan to Share IPD: Yes
upon reasonable request will be provided by the authors